CLINICAL TRIAL: NCT00687024
Title: Determining the Extent of Diffusion Tensor Abnormalities in Focal Cortical Dysplasia
Acronym: FCP
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Charles Raybaud, Division Head, Neuroradiology, The Hospital for Sick Children
Other Study IDs: 1000010634
Record Dates: First submitted 2008-05-26; First posted 2008-05-30 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Focal Cortical Dysplasia; Epilepsy
Keywords: Epilepsy; Magnetic Resonance Imaging; Magnetoencephalography
MeSH Terms: conditions — Focal Cortical Dysplasia; Epilepsy | interventions — Magnetoencephalography; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Magnetoencephalography — MEG will be performed on a whole head Omega 151-channel gradiometer system. At least 15 2-minute periods of spontaneous data are recorded. The sampling rate for data acquisition is 625Hz, with a bandpass filter of 3 to 70 Hz and a notch filter of 60Hz.
Procedure: MR imaging — MR imaging will be performed on a GE 1.5T system using a variety of sequences, including sagittal T1, axial T2, axial FLAIR, coronal dual echo, coronal FLAIR, axial 3D T2 frFSE and axial SPGR.
Procedure: Diffusion Tensor Imaging — Diffusion tensor imaging will be performed on the same scanner, using single shot diffusion-weighted echo planar imaging. Twenty-five 'xial contiguous slices are obtained aligned to the anterior commissure line to cover the whole brain, giving a total imaging time of 4min 40sec.

SUMMARY:
Focal cortical dysplasia (FCD) is a common finding in epilepsy surgery in pediatric patients. Children with intractable epilepsy would have extensive tests to identify the cause of epilepsy; this includes MR brain, video EEG and magnetoencephalography (MEG). The white matter next to FCD is frequently found to be abnormal on pathology. Diffusion tensor imaging (DTI) can be used to study the abnormal white matter and the area that often extends beyond the area that is visible.

DETAILED DESCRIPTION:
Focal cortical dysplasia (FCD) is a highly epileptogenic form of malformation of cortical development that may require surgical resection for epilepsy control. With abnormal development and organization of neurons within the cortex, the white matter projecting from the abnormal cortex is likely to be abnormal as well. The abnormality in the white matter involves not only the subcortical white matter, but also the long tracts in the deep white matter associated with the dysplastic cortex. Histologically, the subcortical white matter adjacent to the dysplastic cortex has been found to be abnormal. Studies using diffusion tensor imaging (DTI) to investigate the white matter adjacent to the MR visible abnormality have demonstrated reduced fractional anisotropy. However, electrographic abnormality in FCD often extends beyond the visible MR abnormality and surgical outcome of epilepsy surgery in FCD is dependent on excising the MR visible abnormality as well as electrographically abnormal area beyond the MR visible abnormality. The cortical and white matter abnormalities are therefore assumed to extend beyond the MR visible lesion. The short-term goal of this study is to determine whether quantitative measures of the abnormal white matter using DTI are able to provide surrogate markers for the extent of FCD. Whilst surgical outcome data is not available for the purpose of this study, these children will be followed up and in the longer term, the extent of FCD as determined by DTI will be compared with clinical outcome post surgery. This study will help determine the potential value of this technique in identifying areas of FCD that appear normal on structural MR. In the long term, this technique can be extended to study children with intractable epilepsy with (i) MR occult lesion and (ii) developmental tumor with MR occult FCD adjacent to the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Children with intractable epilepsy with suspected FCD for MRI & MEG

Exclusion Criteria:

* Children with contraindications to MRI such as those with pacemaker

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with suspected FCD presenting with intractable epilepsy for MRI & MEG. The children will be identified from referral for clinical MRI scans.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the subcortical white matter in the visualized MR abnormality as well as beyond the visualized MR abnormality but subjacent to the MEG dipoles | Immediately after MEG

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raybaud, M.D., Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada